CLINICAL TRIAL: NCT05284825
Title: A Phase II Trial of Intermediate Radiation Dose For Low Grade Follicular Lymphoma
Brief Title: A Phase II Trial of Intermediate Radiation Dose For Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3744
Record Dates: First submitted 2022-03-10; First posted 2022-03-17 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2023-04

CONDITIONS: Follicular Lymphoma
Keywords: radiation
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 12 Gy in 6 daily fractions (Experimental)
  Interventions: Radiation: 12 Gy in 6 daily fractions

INTERVENTIONS:
Radiation: 12 Gy in 6 daily fractions — 12 Gy in 6 daily fractions

SUMMARY:
The purpose of this study is to determine the optimal radiation dose fractionation regimen for low grade follicular lymphoma.

It is hypothesized that the complete response rate with the use of 12 Gy in 6 daily fractions is 80% (10% total width of the confidence interval) at 3 months.

This phase II study will evaluate whether an intermediate dose for follicular lymphoma is associated with excellent response rates while minimizing acute and late toxicity.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years or older
* Pathology review at Sunnybrook Health Sciences Centre showing low grade (grade 1- 2) follicular lymphoma
* Previously un-irradiated stages I-IV low grade follicular lymphoma
* Radiation indicated for local disease control (radical or palliative)
* Able to give informed consent
* Non-bulky targets (less than 7cm)

Exclusion Criteria:

* Systemic therapy (including steroids) for lymphoma within 3 months before or after radiotherapy
* Prognosis less than 3 months
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Complete response within the radiated volume at 1month post radiation | 1 month
  Participants will be assessed for response at 1 month (primary outcome) and then 3 months following completion of radiotherapy, clinically or radiographically, as appropriate.
  Complete response is defined as absence of detectable disease in the radiated volume. Partial response is 50% or more reduction in the volume of disease in the radiated volume. Overall response is defined as complete and partial response. Stable disease is defined as no change in the irradiated tumour or less than 50% reduction. Progressive disease is defined as enlargement of the irradiated tumour

SECONDARY OUTCOMES:
Overall survival, progression-free survival and toxicity | 1 month and 3 month
  Toxicity (6) will be scored according to the Common Terminology Criteria for Adverse Events (CTCAE) definitions (site specific modules), at 1 month and then 3 months following completion of radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: May Tsao, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada